CLINICAL TRIAL: NCT03433963
Title: The Use of L-arginine to Mitigate the Cardiovascular Effects of Exposure to Traffic-related Air Pollution: A Randomized, Double-blind, Placebo-controlled Trial
Brief Title: The Use of L-arginine to Mitigate the Cardiovascular Effects of Exposure to Traffic-related Air Pollution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shaowei Wu, Associate Professor, Peking University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2017074
Record Dates: First submitted 2018-01-31; First posted 2018-02-15 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Blood Pressure; Cardiac Ischemia
Keywords: air pollution; blood pressure; cardiac ischemia; L-arginine; nitric oxide
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-Arg supplement group (Experimental): Study participants in the group will take L-Arg supplement during the trial.
  Interventions: Dietary Supplement: L-Arg supplement
- Control group (Placebo Comparator): Study participants in the group will take placebo during the trial.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: L-Arg supplement — L-Arg supplement will be prepared as pills, administered 9g each day in 3 times for 2 weeks.
  Arms: L-Arg supplement group
Dietary Supplement: Placebo — Placebo will be prepared as pills (the same size, color and shape as of L-Arg), administered 3 times daily for 2 weeks.
  Arms: Control group

SUMMARY:
The present study is aimed to investigate whether oral L-arginine supplementation reduces the adverse cardiovascular effects of exposure to traffic-related air pollution among a group of non-smoking adults with elevated blood pressure.

DETAILED DESCRIPTION:
The present study is designed as a randomized, double-blind, placebo-controlled trial of L-arginine (L-Arg, a precursor of nitric oxide in human body) supplement to counteract the acute cardiovascular effects of exposure to traffic-related air pollution among a group of non-smoking adults with elevated blood pressure. A large number of epidemiological studies have provided compelling evidence that exposure to traffic-related air pollution contributes to the increases in cardiovascular morbidity and mortality, and the mechanism of action includes vasoconstriction and cardiac ischemia. It is well known that nutritional factors are very important determinants of cardiovascular health. However, few studies have explored the joint effects of air pollution and nutritional factors on cardiovascular health. Existing data from many laboratory studies and small clinical trials suggest that L-Arg has beneficial effects on the cardiovascular system by lowering blood pressure and protecting myocardiocytes against external stimuli. The study will explore whether L-Arg supplement improves blood pressure levels and prevents potential cardiac ischemia upon acute exposure to traffic-related air pollution among high-risk individuals.

Dietary intakes, lifestyle habits, use of medication/dietary supplements, blood pressure, resting electrocardiogram and plasma parameters were assessed for potential eligible participants at screening visits. Over 500 participants completed the screening visits, and 118 of them were eligible after a 5-day L-Arg-free run-in period and willing to participate in the following intervention. Eligible participants were assigned to either the interventional group or control group using a computerized method with a randomized block design. They received 2 weeks (may float back and forth for 1-3 days due to scheduling issues) daily doses of either L-Arg (9g/day in 3 times) or placebo and undergo a 2-h exposure scenario (0900-1100 hours) of walking along a traffic road on the 14th day. Participants were counseled to maintain an isocaloric diet and to abstain from other L-Arg rich foods during the study. Concentrations of major traffic-related air pollutants, including particulate matter with an aerodynamic diameter ≤ 2.5 μm (PM2.5), black carbon, and nitrogen dioxide, were measured from the beginning of the 2-h exposure scenario to 22h after exposure or during the 2-h exposure scenario, and primary and secondary outcome measures including blood pressure, ST-segment depression and plasma parameters were assessed repeatedly at various time points (depending on the parameters) around the 2-h exposure scenario. Other environmental factors, including noise, temperature and relative humidity, were also recorded during the 2-h exposure scenario and up to 22h after exposure.

ELIGIBILITY:
Inclusion Criteria:

1. Having elevated systolic blood pressure between 120-160 mmHg, and diastolic blood pressure between 65-100 mmHg, either with or without routine antihypertensive medications.
2. Adults between 50 and 75 years of age, current non-smokers;
3. Do not take routine vasoactive dietary supplements.

Exclusion Criteria:

1. Hypertension with SBP>160 mmHg or DBP>100 mmHg, clinical diagnosis of cardiovascular disease (excluding hypertension), or other important chronic diseases such as coagulopathy, chronic obstructive pulmonary disease, asthma, gastrointestinal diseases, cancer or mental diseases;
2. No routine use of vasoactive dietary supplements,or, if taking, willing to forego their use during the trial.
3. Fasting LDL cholesterol≥4.92 mmol/L or total cholesterol≥6.21 mmol/L or HbA1c>9%;
4. Liver or renal dysfunction;
5. Acute coronary symptoms or unstable clinical manifestations within the past three months;
6. Suffering from allergic diseases/known allergy to ingredients of L-Arg; or those who suffered from acute illness before start of the study;
7. Alcohol or drug addiction;
8. Hepatitis B / hepatitis C virus patient / carrier;
9. History of organ transplants or major surgery in the past year;
10. Exposed to occupational sources of air pollution;
11. Unwilling or unable to provide informed consent or cooperate with all research related procedures.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2019-07-04 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Change in systolic and diastolic blood pressure from before the dietary intervention to before, during, 30min after and 22h after the 2-h exposure scenario | before taking L-Arg supplement/placebo (1st day); before and during the 2-h exposure scenario (14th day); 30min after the exposure scenario (14th day); and 22h after the exposure scenario (15th day).
Change in ST-segment depression from before the dietary intervention to before, during until 22h after the 2-h exposure scenario | before taking L-Arg supplement/placebo (1st day); and 24 hours from the start of 2-h exposure scenario (14th day) until 22h after the exposure scenario (15th day)
Change in ambulatory blood pressure during the 2-h exposure scenario (vs. before the dietary intervention) | during the 2-h exposure scenario (14th day)

SECONDARY OUTCOMES:
Change in plasma L-Arg from before the dietary intervention to before, 30min after and 22h after the 2-h exposure scenario | before taking L-Arg supplement/placebo (1st day); before the 2-h exposure scenario (14th day); 30min after the exposure scenario (14th day); and 22 hours after the exposure scenario (15th day)
Change in plasma nitric oxide (including nitrate and nitrite) from before the dietary intervention to before, 30min after and 22h after the 2-h exposure scenario | before taking L-Arg supplement/placebo (1st day); before the 2-h exposure scenario (14th day); 30min after the exposure scenario (14th day); and 22 hours after the exposure scenario (15th day)
Change in plasma cyclic guanosine monophosphate from before the dietary intervention to before, 30min after and 22h after the 2-h exposure scenario | before taking L-Arg supplement/placebo (1st day); before the 2-h exposure scenario (14th day); 30min after the exposure scenario (14th day); and 22 hours after the exposure scenario (15th day)
Change in plasma C-reactive protein from before the dietary intervention to before, 30min after and 22h after the 2-h exposure scenario | before taking L-Arg supplement/placebo (1st day); before the 2-h exposure scenario (14th day); 30min after the exposure scenario (14th day); and 22 hours after the exposure scenario (15th day)
Change in plasma myeloperoxidase from before the dietary intervention to before, 30min after and 22h after the 2-h exposure scenario | before taking L-Arg supplement/placebo (1st day); before the 2-h exposure scenario (14th day); 30min after the exposure scenario (14th day); and 22 hours after the exposure scenario (15th day)
Change in pulse oxygen saturation from before the dietary intervention to before, 30min after and 22h after the 2-h exposure scenario | before taking L-Arg supplement/placebo (1st day); before the 2-h exposure scenario (14th day); 30min after the exposure scenario (14th day); and 22 hours after the exposure scenario (15th day)
Change in endothelial nitric oxide synthase from before the dietary intervention to before, 30min after and 22h after the 2-h exposure scenario | before taking L-Arg supplement/placebo (1st day); before the 2-h exposure scenario (14th day); 30min after the exposure scenario (14th day); and 22 hours after the exposure scenario (15th day)
Change in two related amino acids (citrulline and ornithine) in L-arg metabolic pathway from before the dietary intervention to before, 30min after and 22h after the 2-h exposure scenario | before taking L-Arg supplement/placebo (1st day); before the 2-h exposure scenario (14th day); 30min after the exposure scenario (14th day); and 22 hours after the exposure scenario (15th day)

CONTACTS AND LOCATIONS:
Overall Officials: Shaowei Wu, PhD, Principal Investigator — Peking University
Locations (3):
- China (3):
  - Qinglongqiao Community Health Service Center, Beijing
  - Malianwa Community Health Service Center, Beijing
  - Shangdi Community Health Service Center, Beijing

IPD SHARING:
Plan to Share IPD: No